CLINICAL TRIAL: NCT04812691
Title: CD19-targeted CAR T Cells （JWCAR029） for Primary Refractory Diffuse Large B Cell Lymphoma, Phase Ⅰ,Open-label,Single-arm,Muticenter Study
Brief Title: CD19-targeted CAR T Cells （JWCAR029） for Primary Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029-003
Record Dates: First submitted 2021-01-18; First posted 2021-03-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Primary refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JWCAR029 (Experimental): The safety and efficacy of JWCAR029 will be evaluated in 1 x 10^8 CAR+T cells dose level
  Interventions: Biological: JWCAR029 (CD19-targeted Chimeric Antigen Receptor Cells)

INTERVENTIONS:
Biological: JWCAR029 (CD19-targeted Chimeric Antigen Receptor Cells) — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JWCAR029. During JWCAR029 production, subjects will receive a conditioning chemotherapy regimen of cyclophosphamide and fludarabine for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive 1 x 10^8 CAR+T cells (JWCAR029) treatment by intravenous (IV) injection.

SUMMARY:
This is a phase I, open-label, single-arm, multicenter study to assess the safety and efficacy of JWCAR029 in adult primary refractory DLBCL subjects in China

DETAILED DESCRIPTION:
This is a phase I, open-label, single-arm, multicenter study conducted in adult subjects with primary refractory DLBCL in China to evaluate the safety, efficacy, pharmacokinetics(PK), pharmacodynamics(PD) of JWCAR029 and collect immune response after JWCAR029 treatment.

One dose level of 1.0 x 10^8 CAR+ T cells is adopted in this study. All sujects will be followed for 2 years after JWCAR029 infusion.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old;
2. Sign on the informed consent;
3. Subject must have histologically confirmed diffuse large B lymphoma and primary refractory with first-line therapy;
4. Subjects have accessible PET-positive lesion and have measurable CT-positive lesion according to Lugano Classification;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
6. Adequate organ function;
7. Adequate vascular access for leukapheresis procedure;
8. Subjects who have previously received CD19 targeted therapy must confirm that lymphoma lesions still express CD19;
9. Women of childbearing potential must agree to use highly effective methods of contraception for 1 year after the last dose of JWCAR029;
10. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method for 1 year after the last dose of JWCAR029

Exclusion Criteria:

1. Subjects who have received second-line treatment or above
2. CD19 negative
3. Primary CNS lymphoma;
4. History of another primary malignancy that has not been in remission for at least 2 years;
5. Subjects has HBV, HCV, HIV or syphilis infection at the time of screening;
6. Deep venous thrombosis (DVT)/Pulmonary embolism (PE), or DVT/PE requires anti-coagulation within 3 months prior to signing the ICF;
7. Subjects with uncontrolled systemic fungal, bacterial, viral or other infection;
8. Presence of acute or chronic graft-versus-host disease (GVHD);
9. History of any serious cardiovascular disease or presence of clinically relevant CNS pathology;
10. Pregnant or nursing women;
11. Subjects using of any chemotherapy, corticisteriod, experiment agents, GVHD therapies, radiation, allo-HSCT or any other therapies for lymphoma must go through a specific wash-out period before leukapheresis;
12. Uncontrolled conditions or unwillingness or inability to follow the procedures required in the protocol;
13. Received CAR T-cell or other genetically-modified T-cell therapy previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Types, frequency, and severity of adverse events and laboratory anomalies | 2 years
  Physiological parameter

SECONDARY OUTCOMES:
Complete response rate (CRR) in primary refractory DLBCL subjects | 1 month
  Investigator evaluated CRR in 1 month
Objective response rate (ORR) in primary refractory DLBCL subjects | 1 month
  Investigator evaluated ORR in 1 month
Best objective response rate (BORR) | 2 years
  The best response from the onset of treatment to the onset of disease progression/recurrence or to the onset of another anticancer treatment
Investigator evaluated CRR | 3 months
  Complete response rate (CRR)
Investigator evaluated ORR (ORR=CR+PR) | 3 months
  Complete response (CR) + partial response（PR）
Duration of response (DOR) | up to 24 months after JWCAR029 infusion
  Time from first response(PR or CR) to disease progression or death from any cause
Duration of complete remission (DoCR) | up to 24 months after JWCAR029 infusion
  Time from complete response (CR) to disease progression or death from any cause
Time to response (TTR) | up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of CR or PR
Time to complete response (TTCR) | up to 24 months after JWCAR029 infusion
  Time from JWCAR029 infusion to first documentation of CR
Pharmacokinetic (PK)- Cmax of JWCAR029 | up to 1 year after JWCAR029 infusion
  Maximum observed concentration of JWCAR029 in peripheral blood
Pharmacokinetic (PK)- Tmax of JWCAR029 | up to 1 year after JWCAR029 infusion
  Time to maximum concentration of JWCAR029 in the peripheral blood
Pharmacokinetic (PK)- AUC of JWCAR029 | up to 1 year after JWCAR029 infusion
  Area under the concentration vs time curve of JWCAR029
Progression-free survival (PFS) | up to 2 year after JWCAR029 infusion
  Progression-free survival
Overall survival (OS) | up to 2 year after JWCAR029 infusion
  Overall survival
Changes of CRP and serum ferritin | 1 year after JWCAR029 infusion
  Changes of inflammation biomarkers-CRP and serum ferritin
Anti-therapeutic JWCAR029 antibody | up to 2 year after JWCAR029 infusion
  The level of anti-therapeutic JWCAR029 antibody after JWCAR029 infusion
The concentration of Car-T cell | up to 2 year after JWCAR029 infusion
  The concentration of Car-T cells
The proportion of Car-T cell subgroups | up to 2 year after JWCAR029 infusion
  The proportion of Car-T cell subgroups after infusion
The concentration of CD19 in tumor biopsy samples | up to 2 year after JWCAR029 infusion
  The concentration of CD19 in tumor biopsy samples
The change of serum cytokines concentration | up to 2 year after JWCAR029 infusion
  The change of serum cytokines concentration after JWCAR029 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Principal Investigator — Ruijin Hospital
Locations (2):
- China (2):
  - Ruijin hospital, Shanghai, Shanghai Municipality
  - Zhejiang university school of medicine first affiliated hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No